CLINICAL TRIAL: NCT05510648
Title: The Effect of High-intensity Laser Therapy in Knee Osteoarthritis
Brief Title: Evaluation of the Effect of High-intensity Laser Therapy in Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Banu Ordahan, Clinical Professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BANU ORDAHAN
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Knee Osteoarthritis; Laser Therapy; Muscle Strength
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity laser therapy (Active Comparator): A total of 15 sessions of hotpack, TENS and exercise program will be applied to the patients for three weeks, 5 days a week, 1 session a day. The hotpack, which is used as a superficial heater, is applied to the knee area for 30 minutes, wrapped in two layers of towels. As analgesic current, conventional TENS is applied to the knee area for 30 minutes with 4 electrodes at 80 Hz frequency, 200 ms current duration. Flow intensity is adjusted according to the patient's tolerance, and the current intensity is increased as the patient's sense of current decreased in the following periods. HILT is applied in analgesic mode for 3 sessions every other day in the first week, and 6 sessions every other day in the biostimulant mode for the next two weeks, for a total of 9 sessions for three weeks.
  Interventions: Other: high-intensity laser therapy; Other: sham high-intensity laser therapy
- Sham high-intensity laser therapy (Sham Comparator): Hotpack, TENS and exercise program applications will be applied to the patients in the same way as in the HILT group, 5 days a week, 1 session a day, a total of 15 sessions for three weeks. HILT is administered as a placebo for three weeks, 3 sessions a week, every other day, for a total of 9 sessions.
  Interventions: Other: high-intensity laser therapy; Other: sham high-intensity laser therapy

INTERVENTIONS:
Other: high-intensity laser therapy — A total of 15 sessions of hotpack, TENS and exercise program will be applied to the patients for three weeks, 5 days a week, 1 session a day. The patients in the HILT group will be treated with a BTL 6000 brand device (Figure 5) for 3 sessions of high-intensity laser with a power of 10.0 w in the first week, energy density of 12 j/cm², every 25 cm² for 2 minutes in analgesic mode, and 5 sessions in the following 2 weeks. While 6 sessions of .0 w power, energy density of 120 j/cm², each 25 cm² for 10 minutes, will be applied in biostimulant mode for 6 sessions for three weeks, is applied in analgesic mode for 3 sessions every other day in the first week, and 6 sessions every other day in the biostimulant mode for the next two weeks, for a total of 9 sessions for three weeks.
Other: sham high-intensity laser therapy — Hotpack, TENS and exercise program applications will be applied to the patients in the same way as in the HILT group, 5 days a week, 1 session a day, a total of 15 sessions for three weeks. HILT is administered as a placebo for three weeks, 3 sessions a week, every other day, for a total of 9 sessions.

SUMMARY:
The aim of this study is to evaluate the effects of high intensity laser therapy (HILT) on range of motion, pain, quality of life, muscle strength and femoral cartilage thickness in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Patients who are admitted and diagnosed with knee osteoarthritis based on anamnesis, physical examination and imaging methods are included in the study.

ELIGIBILITY:
Inclusion Criteria:

1-40-70 years old 2-Diagnosis of knee OA according to ACR clinical and radiological diagnostic criteria 3-Kellgren Lawrence stage II or III 4-Knee pain for at least 6 months 5-Visual analog scale (VAS) score of at least 3 or more

Exclusion Criteria:

1. History of surgery or traumatic injury
2. Inflammatory arthritis
3. History of cancer, bleeding diathesis and psychiatric disease
4. Those who have a disease that limits their participation in exercises (severe chronic obstructive lung disease, severe heart failure, history of cerebrovascular events)
5. Hip and ankle problems
6. Participating in another physical therapy program in the last 3 months
7. History of intra-articular injections in the last 6 months

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-25 (Estimated); Primary Completion 2022-09-25 (Estimated); Study Completion 2022-11-25 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Change from baseline in pain on the VAS at month 3 | Baseline and month 3
  Visual Analog Scale (VAS) is used to measure and monitor the intensity of pain. This is a 10 cm ruler that describes painlessness at one end and the most severe pain at the other. A patient scores his/her pain from 0 to 10.

SECONDARY OUTCOMES:
Knee joint range of motion Change from baseline in knee joint on the measuring the range of motion at knee joint at month 3 | Baseline and month 3
  The range of motion of the patients, consisting of knee flexion and extension, is actively evaluated with a goniometer. In the measurement of the flexion angle, the patient is lying in the prone position and the extension angle is measured as the limitation of extension when the knee joint is at 0 degrees
Femoral cartilage thickness Change from baseline in knee joint on the measuring the femoral cartilage thickness at month 3 | Baseline and month 3
  Femoral cartilage thickness is measured by the same physician by placing the probe axially in the suprapatellar region by ultrasonography while the patient is lying on his back and the knees are in maximum flexion. The distance between the thin hyperechoic line at the synovial cartilage interface and the sharp hyperechoic line at the cartilage-bone interface is defined as cartilage thickness
SF-36 quality of life scale Change from baseline in physical and mental functions on SF-36 quality of life scale at month 3 | Baseline and month 3
  The SF-36 scale measures 8 dimensions of health and consists of 36 items; physical function (10 items), social function (2 items), role related to physical functions limitations (4 items), role limitations due to emotional problems (3 items), mental health (5 items), energy/fatigue (4 items), pain (2 items), and general perception of health (5 items). It is evaluated between 0 and 100 points; 0 represents poor health, 100 represents good health. There are two summary components, the physical component and the mental component
Western OntarioMacMaster (WOMAC) Change from baseline in pain and physical functions on Western OntarioMacMaster scale at month 3 | Baseline and month 3
  It is widely used in studies with knee OA patients. The scale, each question of which is evaluated with a 5-point Likert scale, consists of 24 questions. It is filled by patients. There are pain, physical function and stiffness subscales. Pain subscale is evaluated with five items and is scored between 0-20. The hardness subscale has two items and is scored between 0-8. Function subscale consists of 17 items and is scored between 0-68. A high score indicates poor function, pain or stiffness.
Isokinetic muscle strength measurement Change from baseline in knee joint on the measuring the isokinetic muscle strength at month 3 | Baseline and month 3
  Knee isokinetic muscle strength is measured with the Biodex System-3 isokinetic device . At 60° and 180° angular velocities, the range of motion was 90° flexion 0° extension, after three repetitions at each angular velocity; Measurements are made in a single set-five repetitions with 10 seconds of rest between repetitions

CONTACTS AND LOCATIONS:
Overall Officials: BANU ORDAHAN, Principal Investigator — Meram Medical School, Necmettin Erbakan University, Konya, Turkey